CLINICAL TRIAL: NCT05491226
Title: IIT2021-01-Shiao-CSF1Ri: Reinvigorating TNBC Response to Immunotherapy With Combination Myeloid Inhibition and Radiation
Brief Title: Reinvigorating TNBC Response to Immunotherapy With Combination Myeloid Inhibition and Radiation
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Stephen Shiao (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry); Incyte Corporation (Industry)
Responsible Party: Sponsor-Investigator, Stephen Shiao, Associate Professor, Departments of Radiation Oncology and Biomedical Sciences, Cedars-Sinai Medical Center
Organization: Cedars-Sinai Medical Center (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IIT2021-01-Shiao-CSF1Ri
Record Dates: First submitted 2022-08-04; First posted 2022-08-08 (Actual); Last update posted 2025-08-27 (Actual); Status verified 2025-08

CONDITIONS: TNBC - Triple-Negative Breast Cancer; Breast Cancer
Keywords: pembrolizumab; axatilimab; radiation therapy
MeSH Terms: conditions — Triple Negative Breast Neoplasms; Breast Neoplasms | interventions — pembrolizumab; Radiotherapy; axatilimab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Pembrolizumab with Radiation Therapy and Axatilimab (Experimental)
  Interventions: Drug: Pembrolizumab; Radiation: Radiation Therapy; Drug: Axatilimab

INTERVENTIONS:
Drug: Pembrolizumab — Pembrolizumab 200 mg is administered intravenously at Week 1, then every 3 weeks during the treatment period (6 weeks). Therapy will continue for until initiation of SOC curative-intent treatment (neoadjuvant chemo therapy or surgery) at Week 7.
  Other Names: Keytruda
Radiation: Radiation Therapy — Radiation therapy (RT) consists of 8 Gy for 3 fractions over 3 consecutive days at Week 2.
Drug: Axatilimab — Axatilimab 1 mg/kg is administered intravenously weekly starting 1 week post- RT (Week 3). Therapy will continue until initiation of SOC curative-intent treatment (neoadjuvant chemo therapy or surgery) at Week 7.

SUMMARY:
This is an open-label prospective, single institution, Phase II study of pembrolizumab in combination with radiation therapy and CSF-1R inhibition in patients with high-risk TNBC. The primary objective is to assess the pathologic complete response (pCR) rate where pCR is defined as the absence of invasive disease in the breast and lymph nodes at the time of standard of care (SOC) treatment. Secondary objectives include evaluating the change in tumor infiltrating lymphocytes (TILs), safety and tolerability of the combination, progression-free survival, event-free survival, overall survival, and node clearance.

ELIGIBILITY:
Inclusion Criteria:

* Female patients diagnosed with high-risk triple negative breast cancer (TNBC) with intent for neoadjuvant therapy.
* Low tumor-infiltrating lymphocyte (TIL) score, defined as stromal TIL (sTIL) ≤40%; or node-positive; or combined positive score (CPS) < 10 or PD-L1 tumor positivity <1%.
* Written informed consent obtained from subject and ability for subject to comply with the requirements of the study, including consent for research blood draws and use of available archived tissue.
* Age ≥ 18 years of age on day of signing informed consent.
* Histologically or cytologically-confirmed TNBC (defined as ER <1%, PR<1%, her-2-neu 0-1+ by IHC or FISH-negative).
* If an archived tumor tissue is unavailable, be willing to provide tissue from a newly obtained core or excisional biopsy of a tumor lesion. Newly-obtained is defined as a specimen obtained up to 6 weeks (42 days) prior to initiation of treatment on Day 1 of RT.
* Have a performance status of 0 or 1 on the ECOG Performance Scale.
* Demonstrate adequate organ function.
* Female subject of childbearing potential should have a negative serum or urine pregnancy test or documentation of absence of pregnancy by a gynecologist within 14 days of initiating first dose of pembrolizumab (1 week lead-in) for eligibility verification.
* Female subjects of childbearing potential should be willing to comply to the contraceptive guidance in Appendix 12.2 during the treatment period through 120 days after the last dose of study medication. Subjects of childbearing potential are those who have not been surgically sterilized or have not been free from menses for > 1 year.

Exclusion Criteria:

* Evidence of metastatic disease.
* Has received prior radiotherapy within 2 weeks of start of study intervention.
* Is currently participating and receiving study therapy or has participated in a study of an investigational agent and received study therapy or used an investigational device within 4 weeks of the first dose of treatment.
* Has a diagnosis of immunodeficiency or is receiving systemic steroid therapy or any other form of immunosuppressive therapy within 7 days prior to the first dose of trial treatment.
* Has a known history of active TB (Bacillus Tuberculosis).
* Hypersensitivity to pembrolizumab or any of its excipients.
* Has had a prior anti-cancer monoclonal antibody (mAb) within 4 weeks prior to study Day 1 or who has not recovered (i.e., > Grade 1 or at baseline) from adverse events due to agents administered more than 4 weeks earlier.
* Has had prior chemotherapy or targeted small molecule therapy within 2 weeks prior to study Day 1 or who has not recovered (i.e., > Grade 1 or at baseline) from adverse events due to a previously administered agent. Note: Subjects with ≤ Grade 2 neuropathy are an exception to this criterion and may qualify for the study.
* Has a known additional malignancy that progressed or required treatment in the last 5 years. Exceptions include basal cell carcinoma of the skin or squamous cell carcinoma of the skin that has undergone potentially curative therapy or in situ cervical cancer.
* Has known active central nervous system (CNS) metastases and/or carcinomatous meningitis. Subjects with previously treated brain parenchymal metastases may participate provided they are stable (without evidence of progression by imaging for at least four weeks prior to the first dose of trial treatment and any neurologic symptoms have returned to baseline), have no evidence of new or enlarging brain metastases, and are not using steroids for at least 7 days prior to trial treatment. This exception does not include carcinomatous meningitis, which is excluded regardless of clinical stability.
* Has active autoimmune disease that has required systemic treatment in the past 2 years (i.e. with use of disease modifying agents, corticosteroids or immunosuppressive drugs). Replacement therapy (e.g., thyroxine, insulin, or physiologic corticosteroid replacement therapy for adrenal or pituitary insufficiency, etc.) is not considered a form of systemic treatment.
* Has known history of/active, non-infectious pneumonitis requiring treatment with steroids or has history of/active interstitial lung disease.
* Has an active infection requiring systemic therapy.
* Has a history or current evidence of any condition, therapy, or laboratory abnormality that might confound the results of the trial, interfere with the subject's participation for the full duration of the trial, or is not in the best interest of the subject to participate, in the opinion of the treating investigator.
* Has known psychiatric or substance abuse disorders that would interfere with cooperation with the requirements of the trial.
* Is pregnant or breastfeeding, or expecting to conceive within the projected duration of the trial, starting with the pre-screening or screening visit through 120 days after the last dose of trial treatment. A WOCBP who has a positive urine pregnancy test within 2 weeks prior to start of study treatment (first dose of pembrolizumab). If the urine test is positive or cannot be confirmed as negative, a serum pregnancy test will be required. Note: Negative urine or serum pregnancy test is also conducted within 72 hours prior to C1D1 for study procedures but if screening pregnancy test is done within 72 hours of C1D1, it is not required to be repeated..
* Has a known history of Human Immunodeficiency Virus (HIV) (HIV 1/2 antibodies).
* Has a known history of active Hepatitis B (e.g., HBsAg reactive) or known active Hepatitis C (e.g., HCV RNA [qualitative] is detected).
* Has received a live vaccine or live-attenuated vaccine within 30 days of planned start of pembrolizumab. Administration of killed vaccines is allowed.
* Has had an allogenic tissue/solid organ transplant.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Estimated)
Dates: Start 2023-11-17 (Actual); Primary Completion 2026-12-01 (Estimated); Study Completion 2026-12-01 (Estimated)

PRIMARY OUTCOMES:
Pathological complete response (pCR) rate. | From treatment start date until the time of curative-intent treatment, approximately 7 weeks.
  The proportion of patients with absence of invasive disease in the breast and lymph nodes at the time of SOC curative-intent treatment.

SECONDARY OUTCOMES:
Change in tumor-infiltrating lymphocytes (TILs) from biopsies. | From Week 1 and at the time of SOC curative-intent treatment, approximately 7 weeks from start of trial treatment..
  An increase in the tumor-infiltrating lymphocyte score as measured by Salgado criteria, is an indicator of immune system engagement.
Number of adverse events related to study treatment (pembrolizumab with radiation and axatilimab). | From start of treatment until 1 year post-treatment.
  Adverse events are graded per NCI CTCAE v.5
Event-free survival (EFS). | Assessed up to 3 years.
  The length of time from the start of study treatment to the first occurrence of recurrent disease, or death due to breast cancer.
Overall Survival (OS). | From C1D1 until death, up to 3 years after end of study treatment.
  Assessed from the start of study treatment until death due to any cause.
Node clearance. | From C1D1 until EOT, approximately 7 weeks.
  Assessed by the proportion of node-positive patients who become node-negative post study treatment (by EOT).

CONTACTS AND LOCATIONS:
Overall Officials: Stephen L Shiao, MD, PhD, Principal Investigator — CSMC
Locations (1):
- Cedars-Sinai Medical Center, Los Angeles, California, United States

IPD SHARING:
Plan to Share IPD: No